CLINICAL TRIAL: NCT04396054
Title: Comparison of Double Y-shaped Plates and Lag Screws in Fixation of Anterior Mandibular Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lydia Nabil (Other)
Responsible Party: Sponsor-Investigator, Lydia Nabil, Assistant Professor of Oral and Maxillofacial Surgery, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAlexandriaDentSurg1
Record Dates: First submitted 2020-05-09; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lag Screws (Active Comparator): Group 1: underwent open reduction and internal fixation using two lag screws.
  Interventions: Device: Lag Screws
- Double Y-shaped plates (Active Comparator): Group 2: underwent open reduction and internal fixation using double Y-shaped plates.
  Interventions: Device: double Y-shaped plates

INTERVENTIONS:
Device: Lag Screws — Method of internal fixation
  Arms: Lag Screws
Device: double Y-shaped plates — Method of internal fixation
  Arms: Double Y-shaped plates

SUMMARY:
This study is a prospective randomized controlled clinical trial. It was performed on sixteen patients with anterior mandibular fractures, to compare Double Y-shaped plates and Lag Screws in fracture fixation from clinical and radiographic perspectives.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled clinical trial. It was performed on sixteen patients with anterior mandibular fractures, selected from those admitted to the Emergency Department of Alexandria University Hospital. Ethical approval for the study was obtained from the regional Ethical Review Board of the Faculty of Dentistry, Alexandria University. A written informed consent was signed by patients before the operation.

Patients were divided equally into two groups, each consisting of eight patients. Assignment of each patient into one of either group was done using computer random numbers.

Group 1: underwent open reduction and internal fixation using two lag screws. Group 2: underwent open reduction and internal fixation using double Y-shaped plates.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* with age ranging from 25 to 45 years,
* suffering from anterior fractures of the mandible (symphyseal or parasymphyseal)

Exclusion Criteria:

* old fractures,
* infected fractures
* comminuted fractures

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
progress of fracture healing in the postoperative period | after 6 months
  Measurement of bone density in the fracture line using CBCT at 6 points and calculation of mean bone density
Sensory nerve function using dental probe to assess sensory changes along mental nerve distribution and comparing it to the contralateral side | up to 6 months
  Detection of nerve injury by examining sensory nerve function using dental probe to assess sensory changes along mental nerve distribution and comparing it to the contralateral side

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No